CLINICAL TRIAL: NCT03166332
Title: Improving Mothers for a Better PrenAtal Care Trial Barcelona
Acronym: IMPACTBCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Eduard Gratacós Solsona, Director of ICGON and BCNatal, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMPACT BCN
Record Dates: First submitted 2017-04-19; First posted 2017-05-25 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Intrauterine Growth Restriction; Fetal Growth Retardation
Keywords: Mindfulness; Mediterranean diet; Neurodevelopment; Epigenetics; Fetal growth restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Diet, Mediterranean; Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 3 arms of intervention
Who Masked: Care Provider
Masking Description: Care provider will not know the arm of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean diet (Active Comparator): Mediterranean diet supplemented with extra-virgin olive oil and mixed nuts.
  Interventions: Behavioral: Mediterranean diet
- Mindfulness (Active Comparator): Mindfulness-Based Stress Reduction program (MBSR)
  Interventions: Behavioral: Mindfulness
- No intervention (No Intervention): No intervention strategy

INTERVENTIONS:
Behavioral: Mediterranean diet — Mediterranean diet supplemented with extra-virgin olive oil and nuts
  Arms: Mediterranean diet
Behavioral: Mindfulness — Mindfulness-Based Stress Reduction program (MBSR)
  Arms: Mindfulness

SUMMARY:
High risk women for growth restricted fetuses will randomized in the second trimester into different strategies applied to the mothers: a stress reduction program based on mindfulness techniques or a nutrition interventional program based on Mediterranean diet.

DETAILED DESCRIPTION:
Randomized controlled trial among women at higher risk to have a growth restricted fetus (30%) according to Royal College of Obstetrics and Gynecology (RCOG) Guidelines. These high-risk women will be randomized in order to evaluate an improvement in several outcomes thanks to different strategies applied to the mothers: a stress reduction program based on mindfulness techniques or a nutrition interventional program based on Mediterranean diet.

Main hypothesis: specific interventions improving maternal lifestyle and well being have a positive impact on pregnancy outcomes as well as on fetal growth and development.

Secondary hypothesis is that interventions to improve maternal lifestyle well being have a positive impact on offspring's outcome later in life, in terms of neurodevelopment and cardiovascular profile, mediated by epigenetic changes in offspring.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age at recruitment ≥18 years
* Speak Spanish fluently
* Viable singleton non-malformed fetus
* High-risk pregnancy to develop FGR.
* 19-23 weeks of gestation

Exclusion Criteria:

* Fetal anomalies including chromosomal abnormalities or structural malformations detected by ultrasound.
* Mental retardation or other mental or psychiatric disorders that impose doubts regarding the true patient´s willingness to participate in the study.
* No possibility to come to additional visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1221 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fetal Growth Restriction (FGR) | Delivery
  Birth weight <10th percentile

SECONDARY OUTCOMES:
Adverse Perinatal Outcome (APO) Adverse Perinatal Outcome (APO) | Pregnancy
  Development of one of the following conditions: preeclampsia, preterm delivery, severe FGR (birth weight <3rd percentile), perinatal mortality, metabolic acidosis, mejor neonatal morbidity (presence of intraventricular hemorrhage grade III/IV, necrotizing enterocolitis, periventricular leucomalacia, sepsis, broncopulmonary dysplasia, hypoxic ischemic encephalopathy)

OTHER OUTCOMES:
Fetal Programming | Up to 24 months of age
  Neurodevelopment assessment with Bayley III test
Epigenetics | Delivery
  Different epigenetic changes in fetal cord blood in pregnancies affected by FGR who attend the interventional program as compared to pregnancies with no intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Sant Joan de Deu, Barcelona

IPD SHARING:
Plan to Share IPD: No
Participants will be recruited in our unit and data will be available only for researchers involved in the study.

REFERENCES:
- [Derived] Selma-Royo M, Crispi F, Castro-Barquero S, Casas I, Larroya M, Genero M, Paules C, Benitez L, Youssef L, Pascal R, Encabo N, Nakaki A, Martin-Asuero A, Oller-Guzman MT, Arranz A, Vieta E, Casas R, Estruch R, Gratacos E, Collado MC, Crovetto F. Effects of Mediterranean diet or Mindfulness-Based Stress Reduction during pregnancy on maternal gut and vaginal microbiota: a subanalysis of the Improving Mothers for a better PrenAtal Care Trial BarCeloNa (IMPACT BCN) trial. Am J Clin Nutr. 2025 Oct;122(4):1121-1133. doi: 10.1016/j.ajcnut.2025.07.030. Epub 2025 Aug 5. PMID 40759394
- [Derived] Castro-Barquero S, Crovetto F, Estruch R, Ruiz-Leon AM, Larroya M, Sacanella E, Casanovas-Garriga F, Casas I, Nakaki A, Youssef L, Trejo-Dominguez A, Benitez L, Genero M, Vieta E, Gratacos E, Crispi F, Casas R. Validation of a pregnancy-adapted Mediterranean Diet Adherence Screener (preg-MEDAS): a validation study nested in the Improving Mothers for a better PrenAtal Care Trial BarCeloNa (IMPACT BCN) trial. Am J Clin Nutr. 2024 Aug;120(2):449-458. doi: 10.1016/j.ajcnut.2024.05.025. Epub 2024 Jun 1. PMID 38830408
- [Derived] Nakaki A, Crovetto F, Urru A, Piella G, Borras R, Comte V, Vellve K, Paules C, Segales L, Dacal M, Gomez Y, Youssef L, Casas R, Castro-Barquero S, Martin-Asuero A, Oller Guzman T, Morilla I, Martinez-Aran A, Camacho A, Pascual Tutusaus M, Arranz A, Rebollo-Polo M, Gomez-Chiari M, Bargallo N, Pozo OJ, Gomez-Gomez A, Izquierdo Renau M, Eixarch E, Vieta E, Estruch R, Crispi F, Gonzalez-Ballester MA, Gratacos E. Effects of Mediterranean diet or mindfulness-based stress reduction on fetal and neonatal brain development: a secondary analysis of a randomized clinical trial. Am J Obstet Gynecol MFM. 2023 Dec;5(12):101188. doi: 10.1016/j.ajogmf.2023.101188. Epub 2023 Oct 14. PMID 37839546
- [Derived] Crovetto F, Nakaki A, Arranz A, Borras R, Vellve K, Paules C, Boutet ML, Castro-Barquero S, Freitas T, Casas R, Martin-Asuero A, Oller Guzman T, Morilla I, Martinez-Aran A, Camacho A, Pasqual M, Izquierdo Renau M, Pozo OJ, Gomez-Gomez A, Estruch R, Vieta E, Crispi F, Gratacos E. Effect of a Mediterranean Diet or Mindfulness-Based Stress Reduction During Pregnancy on Child Neurodevelopment: A Prespecified Analysis of the IMPACT BCN Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2330255. doi: 10.1001/jamanetworkopen.2023.30255. PMID 37606923
- [Derived] Crovetto F, Crispi F, Casas R, Martin-Asuero A, Borras R, Vieta E, Estruch R, Gratacos E; IMPACT BCN Trial Investigators. Effects of Mediterranean Diet or Mindfulness-Based Stress Reduction on Prevention of Small-for-Gestational Age Birth Weights in Newborns Born to At-Risk Pregnant Individuals: The IMPACT BCN Randomized Clinical Trial. JAMA. 2021 Dec 7;326(21):2150-2160. doi: 10.1001/jama.2021.20178. PMID 34874420
- [Derived] Crovetto F, Crispi F, Borras R, Paules C, Casas R, Martin-Asuero A, Arranz A, Vieta E, Estruch R, Gratacos E. Mediterranean diet, Mindfulness-Based Stress Reduction and usual care during pregnancy for reducing fetal growth restriction and adverse perinatal outcomes: IMPACT BCN (Improving Mothers for a better PrenAtal Care Trial BarCeloNa): a study protocol for a randomized controlled trial. Trials. 2021 May 24;22(1):362. doi: 10.1186/s13063-021-05309-2. PMID 34030703